CLINICAL TRIAL: NCT01208025
Title: The Assessment of the Plaque at RISK by Non-invasive (Molecular) Imaging and Modelling (ParisK): Prospective Clinical Study for Diagnosis Efficacy for High Risk Plaque and Stroke.
Brief Title: ParisK: Validation of Imaging Techniques
Acronym: ParisK
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-2-082
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2016-09

CONDITIONS: Stroke; Atherosclerosis
Keywords: Plaque; Imaging
MeSH Terms: conditions — Stroke; Atherosclerosis; Plaque, Amyloid | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- symptomatic carotid stenosis 30-69%: Patients with neurological symptoms due to ischemia in the carotid artery territory and with a carotid stenosis between 30% and 69% according to the European Carotid Surgery Trial (ECST) criteria.
  Interventions: Other: Magnetic Resonance Imaging (MRI), Multidetector Computed Tomography (MDCT), Ultrasonography (US), Transcranial Doppler (TCD)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI), Multidetector Computed Tomography (MDCT), Ultrasonography (US), Transcranial Doppler (TCD) — 3 Tesla Magnetic Resonance Imaging (MRI), Multidetector Computed Tomography (MDCT), Ultrasonography (US), Transcranial Doppler (TCD)

SUMMARY:
The possibility of the identification of the risk of rupture of a carotid plaque will have tremendous impact in clinical decision making. Firstly, in symptomatic patients with a 30-69% stenosis, who are currently not operated upon according to the current guidelines, identification of the risk of rupture plaque could identify patients who have a high risk of recurrent stroke, and would benefit of carotid intervention, such as endarterectomy or stent placement. This could potentially prevent a substantial number of strokes. Secondly, in all symptomatic patients with a 70-99% stenosis carotid intervention should be considered, according to the guidelines. However, only one out of six patients with a 70-99% stenosis benefits from a carotid intervention. Identification of patients with a high risk of a recurrent stroke would reduce the number of unnecessary interventions substantially.

The main objective is to show whether imaging characteristics assessed at baseline can predict clinical events in patients with a 30-69 % symptomatic carotid stenosis.

ELIGIBILITY:
Inclusion Criteria:

* neurological symptoms due to ischemia in the carotid artery territory as diagnosed by their neurologist based on anamneses, physical examination and brain imaging (CT or MRI)
* carotid artery stenosis < 70% (upper cut-off value is based on the NASCET criteria, the lower cut-off value is an atherosclerotic plaque with a thickness of at least 2-3 mm, which corresponds to an ECST stenosis of 30%
* written informed consent

Exclusion Criteria:

* patients with probable cardiac source of embolism (rhythm disorders, mitral valve stenosis, prolapse or calcification, mechanical cardiac valves, recent myocardial infarction, left ventricular thrombus, atrial myxoma, endocarditis, dilated cardiomyopathy, patent foramen ovale) or a clotting disorder
* patients with evident other cause of neurological symptoms than carotid stenosis due to atherosclerotic disease (like demyelinating diseases, epilepsy, congenital brain disorders, aneurysms, fibromuscular dysplasia etc)
* patients already scheduled for carotid endarterectomy or stenting.
* severe co-morbidity, dementia or pregnancy
* standard contra-indications for MRI
* patients who have a documented allergy to MRI or CT contrast media
* patients with renal clearance < 30 ml/minute are not eligible to undergo contrast-enhanced MRI
* patients with renal clearance < 60 ml/minute are not eligible to undergo MDCT
* patients who had a TIA or minor stroke more than 3 months before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurological symptoms due to ischemia in the carotid artery territory and with a carotid stenosis between 30-69% according to the ECST criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2010-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
stroke | within 5 years of follow-up
  Ipsilateral recurrent ischemic stroke, transient ischaemic attack (TIA) or new ischemic brain lesions on follow-up brain MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Eline Kooi, PhD, Principal Investigator — Maastricht University Medical Center
Locations (4):
- Netherlands (4):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Academic Medical Center, Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Tziotziou A, Liu Y, Fontana F, Bierens J, Nederkoorn PJ, de Jong PA, Kooi ME, Mess W, van der Lugt A, van der Steen AFW, Bos D, Wentzel JJ, Akyildiz AC. Pressure- and flow-driven biomechanical factors associate with carotid atherosclerosis assessed by computed tomography angiography. Atherosclerosis. 2025 Sep;408:120415. doi: 10.1016/j.atherosclerosis.2025.120415. Epub 2025 Jun 26. PMID 40617722
- [Derived] Kassem M, Gorissen T, Albenwan M, Bierens J, van Dam-Nolen DHK, Liem MI, Hofman PAM, Wildberger JE, Hendrikse J, Mess W, Nederkoorn PJ, Bos D, Nelemans P, van Oostenbrugge RJ, Kooi ME. The relationship between fibrous cap status or plaque surface morphology and intraplaque hemorrhage volume over time: The PARISK Study. J Stroke Cerebrovasc Dis. 2025 May;34(5):108283. doi: 10.1016/j.jstrokecerebrovasdis.2025.108283. Epub 2025 Mar 12. PMID 40081118
- [Derived] Aizaz M, Bierens J, Gijbels MJJ, Schreuder THCML, van Orshoven NP, Daemen JHC, Mess WH, Flohr T, van Oostenbrugge RJ, Postma AA, Kooi ME. Differentiation of Atherosclerotic Carotid Plaque Components With Dual-Energy Computed Tomography. Invest Radiol. 2025 Aug 1;60(8):508-516. doi: 10.1097/RLI.0000000000001153. Epub 2025 Jan 22. PMID 39836610
- [Derived] Nies KPH, Aizaz M, van Dam-Nolen DHK, Goring TCD, Schreuder TAHCML, van Orshoven NP, Postma AA, Bos D, Hendrikse J, Nederkoorn P, van der Geest R, van Oostenbrugge RJ, Mess WH, Kooi ME. Signal intensity and volume of carotid intraplaque hemorrhage on magnetic resonance imaging and the risk of ipsilateral cerebrovascular events: The Plaque At RISK (PARISK) study. J Cardiovasc Magn Reson. 2024 Winter;26(2):101049. doi: 10.1016/j.jocmr.2024.101049. Epub 2024 Jun 13. PMID 38878969
- [Derived] van Dam-Nolen DHK, Truijman MTB, van der Kolk AG, Liem MI, Schreuder FHBM, Boersma E, Daemen MJAP, Mess WH, van Oostenbrugge RJ, van der Steen AFW, Bos D, Koudstaal PJ, Nederkoorn PJ, Hendrikse J, van der Lugt A, Kooi ME; PARISK Study Group. Carotid Plaque Characteristics Predict Recurrent Ischemic Stroke and TIA: The PARISK (Plaque At RISK) Study. JACC Cardiovasc Imaging. 2022 Oct;15(10):1715-1726. doi: 10.1016/j.jcmg.2022.04.003. Epub 2022 Jun 15. PMID 36202450
- [Derived] van Dam-Nolen DHK, van Egmond NCM, Dilba K, Nies K, van der Kolk AG, Liem MI, Kooi ME, Hendrikse J, Nederkoorn PJ, Koudstaal PJ, van der Lugt A, Bos D. Sex Differences in Plaque Composition and Morphology Among Symptomatic Patients With Mild-to-Moderate Carotid Artery Stenosis. Stroke. 2022 Feb;53(2):370-378. doi: 10.1161/STROKEAHA.121.036564. Epub 2022 Jan 5. PMID 34983237
- [Derived] Crombag GAJC, van Hoof RHM, Holtackers RJ, Schreuder FHBM, Truijman MTB, Schreuder TAHCML, van Orshoven NP, Mess WH, Hofman PAM, van Oostenbrugge RJ, Wildberger JE, Kooi ME. Symptomatic Carotid Plaques Demonstrate Less Leaky Plaque Microvasculature Compared With the Contralateral Side: A Dynamic Contrast-Enhanced Magnetic Resonance Imaging Study. J Am Heart Assoc. 2019 Apr 16;8(8):e011832. doi: 10.1161/JAHA.118.011832. PMID 30971168
- [Derived] van Dijk AC, Donkel SJ, Zadi T, Sonneveld MAH, Schreuder FHBM, Chohan MF, Koudstaal PJ, Leebeek FWG, Saxena R, Hendrikse J, Kooi ME, van der Lugt A, de Maat MPM. Association between fibrinogen and fibrinogen gamma' and atherosclerotic plaque morphology and composition in symptomatic carotid artery stenosis: Plaque-At-RISK study. Thromb Res. 2019 May;177:130-135. doi: 10.1016/j.thromres.2019.02.030. Epub 2019 Feb 27. PMID 30897531
- [Derived] Crombag GAJC, Schreuder FHBM, van Hoof RHM, Truijman MTB, Wijnen NJA, Voo SA, Nelemans PJ, Heeneman S, Nederkoorn PJ, Daemen JH, Daemen MJAP, Mess WH, Wildberger JE, van Oostenbrugge RJ, Kooi ME. Microvasculature and intraplaque hemorrhage in atherosclerotic carotid lesions: a cardiovascular magnetic resonance imaging study. J Cardiovasc Magn Reson. 2019 Mar 4;21(1):15. doi: 10.1186/s12968-019-0524-9. PMID 30832656
- [Derived] Steinbuch J, van Dijk AC, Schreuder F, Truijman M, Hendrikse J, Nederkoorn PJ, van der Lugt A, Hermeling E, Hoeks A, Mess WH. Definition of common carotid wall thickness affects risk classification in relation to degree of internal carotid artery stenosis: the Plaque At RISK (PARISK) study. Cardiovasc Ultrasound. 2017 Apr 4;15(1):9. doi: 10.1186/s12947-017-0097-4. PMID 28376791
- [Derived] de Rotte AA, Truijman MT, van Dijk AC, Liem MI, Schreuder FH, van der Kolk AG, de Kruijk JR, Daemen MJ, van der Steen AF, de Borst GJ, Luijten PR, Nederkoorn PJ, Kooi ME, van der Lugt A, Hendrikse J. Plaque components in symptomatic moderately stenosed carotid arteries related to cerebral infarcts: the plaque at RISK study. Stroke. 2015 Feb;46(2):568-71. doi: 10.1161/STROKEAHA.114.008121. Epub 2015 Jan 6. PMID 25563640